CLINICAL TRIAL: NCT03811028
Title: An Open, Single-arm, Multicenter Extension Study to Assess the Safety, Tolerability, and Efficacy of Long-term SOBI003 Treatment in Pediatric MPS IIIA Patients
Brief Title: A Study to Assess the Safety, Tolerability, and Efficacy of Long-term SOBI003 Treatment in Pediatric MPS IIIA Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOBI003-002
Record Dates: First submitted 2018-12-17; First posted 2019-01-22 (Actual); Results first posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2021-12

CONDITIONS: Sanfilippo Syndrome Type A (MPS IIIA)
MeSH Terms: conditions — Mucopolysaccharidosis III

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SOBI003 (Experimental): SOBI003 solution, 20 mg/mL, is mixed with NaCl 0.9% infusion solution prior to administration. For a bodyweight < 25 kg, the total infusion volume is 100 mL. For a bodyweight ≥ 25 kg, the total infusion volume is 250 mL.
  SOBI003 is administered as i.v. infusions given once weekly for a duration of 80 weeks (from Week 25 until Week 104 following the first 24 weeks of SOBI003 administration in the FIH study (SOBI003-001) study. The SOBI003 dose will be adjusted to the highest dose that has been declared safe by the safety review committee on the FIH study.Hence, dose adjustments may occur a couple of times on the extension study until the final decided dose has been determined.
  Interventions: Drug: SOBI003

INTERVENTIONS:
Drug: SOBI003 — weekly i.v. infusion
  Other Names: Modified recombinant human sulphamidase

SUMMARY:
MPS IIIA, also known as Sanfilippo A, is an inherited lysosomal storage disease (LSD). MPS IIIA is caused by a deficiency in sulfamidase, one of the enzymes involved in the lysosomal degradation of the glycosaminoglycan (GAG) heparan sulfate (HS). The natural course of MPS IIIA is characterized by devastating neurodegeneration with initially mild somatic involvement. The aim of the present study is to assess the safety, tolerability and efficacy of long-term SOBI003 treatment. SOBI003 is a chemically modified recombinant human (rh) Sulfamidase developed as an enzyme replacement therapy (ERT).

DETAILED DESCRIPTION:
This is an open, single-arm, multicenter extension study to assess the safety, tolerability and efficacy of long-term SOBI003 treatment in pediatric MPS IIIA patients. The study is an extension of the First in Human (FIH) SOBI003-001 study, allowing continuous treatment of SOBI003 for up to 2 years. Study patients who complete Week 24 of the FIH study (SOBI003-001) will be invited to continue to Week 25 in the extension study.

When entering the extension study, these patients will receive the highest dose that has been declared safe in the ongoing FIH study (SOBI003-001). Upon completion of the FIH study, an analysis aimed at selecting the dose for forthcoming studies will take place. Once the dose has been selected, this dose will be applied to all patients enrolled in the extension study. The total duration of the extension study for an individual patient is 80 weeks, resulting in a total of 104 weeks (2 years) of SOBI003 treatment.

ELIGIBILITY:
Inclusion Criteria:

* Completion of study SOBI003-001
* Informed consent obtained from the patient´s legally authorized representative

Exclusion Criteria:

* If, in the opinion of the investigator, there are patient specific safety concerns that contraindicates further treatment with SOBI003

Ages: 18 Months to 78 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2019-01-19 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Harmatz, MD, Principal Investigator — Children´s Hospital and Research Center, Oakland
Locations (3):
- United States (2):
  - Children´s Hospital and research center, Oakland, California
  - University of North Carolina hospitals, Chapel Hill, North Carolina
- Gazi University Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harmatz P, Muenzer J, Ezgu F, Dalen P, Huledal G, Lindqvist D, Gelius SS, Wiken M, Onnestam K, Broijersen A. Chemically modified recombinant human sulfamidase (SOBI003) in mucopolysaccharidosis IIIA patients: Results from an open, non-controlled, multicenter study. Mol Genet Metab. 2022 Aug;136(4):249-259. doi: 10.1016/j.ymgme.2022.06.008. Epub 2022 Jun 28. PMID 35835061

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Group 1: SOBI003 initial dose 3 mg/kg, once weekly from infusion week 25 to week 104
  SOBI003: weekly i.v. infusion
- Dose Group 2: SOBI003 initial dose 10 mg/kg, once weekly from infusion week 25 to week 104
  SOBI003: weekly i.v. infusion
Period: Overall Study
Arm/Group | Dose Group 1 | Dose Group 2
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Group 1 | Dose Group 2 | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: months] | 52.0 (23.8) | 34.7 (12.7) | 43.3 (19.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety as Measured by Adverse Events Frequencies (by Type and Severity)
Description: Number of adverse events, by type and severity, from week 25 up to week 104
Time Frame: From infusion week 25 up to week 104
Measure: Number; unit: events
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
events
  Any adverse event | 174 | 355
  Any non-treatment emergent serious adverse event | 0 | 1
  Any treatment emergent adverse event (TEAE) | 174 | 351
  Any drug-related TEAE | 69 | 202
  Any non-serious TEAE | 172 | 342
  Any serious TEAE | 2 | 9
  Any serious drug-related TEAE | 0 | 0
  Any TEAE leading to study and/or treatment withdrawal | 0 | 0
  Any drug-related TEAE leading to study and/or treatment withdrawal | 0 | 0
  Any serious TEAE leading to study and/or treatment withdrawal | 0 | 0
  Any TEAE leading to death | 0 | 0
  Any Infusion Related Reaction | 46 | 78

2. Secondary Outcome: The Observed SOBI003 Serum Concentration Immediately Before the Start of Infusion of SOBI003
Description: The observed SOBI003 serum concentration immediately before the start of infusion of SOBI003 (CPre-dose) Blood samples for serum PK analysis were collected either by centrally (i.e., using a catheter in the central venous port) or peripheral (i.e., by venipuncture). Central venous sampling is more convenient than repeated venipuncture.
Time Frame: Weeks 38, 52, 78 and 104
Population: The table report number of available pharmacokinetic (PK) samples
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
ng/mL
  Week 38 - central serum: number analyzed (Participants) | 0 | 1
  Week 38 - central serum |  | 120.0 (NA) — Only one sample analyzed
  Week 52 - central serum: number analyzed (Participants) | 0 | 0
  Week 78 - central serum: number analyzed (Participants) | 1 | 1
  Week 78 - central serum | 47.0 (NA) — Only one sample analyzed | 75.0 (NA) — Only one sample analyzed
  Week 104 - central serum: number analyzed (Participants) | 1 | 0
  Week 104 - central serum | 2610 (NA) — Only one sample analyzed |
  Week 38 - peripheral serum: number analyzed (Participants) | 1 | 2
  Week 38 - peripheral serum | 49 (NA) — Only one sample analyzed | 30 (14.142)
  Week 52 - peripheral serum: number analyzed (Participants) | 1 | 2
  Week 52 - peripheral serum | 123 (NA) — Only one sample analyzed | 11770 (16312)
  Week 78 - peripheral serum: number analyzed (Participants) | 2 | 0
  Week 78 - peripheral serum | 208.5 (234.05) |
  Week 104 - peripheral serum: number analyzed (Participants) | 2 | 3
  Week 104 - peripheral serum | 765.5 (125.16) | 66.33 (49.571)

3. Secondary Outcome: The Observed SOBI003 Serum Concentration at the End of Infusion of SOBI003
Description: The observed SOBI003 serum concentration at the end of infusion of SOBI003 (CEnd of inf) Blood samples for serum PK analysis were collected either by centrally (i.e., using a catheter in the central venous port) or peripheral (i.e., by venipuncture). Central venous sampling is more convenient than repeated venipuncture.
Time Frame: Weeks 38, 52, 78 and 104
Population: The table report number of available pharmacokinetic (PK) samples
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
ng/mL
  Week 38 - central serum: number analyzed (Participants) | 0 | 1
  Week 38 - central serum |  | 210000 (NA) — Only one sample analyzed
  Week 38 - peripheral serum: number analyzed (Participants) | 3 | 2
  Week 38 - peripheral serum | 14370 (14583) | 109500 (3535.5)
  Week 52 - central serum: number analyzed (Participants) | 1 | 1
  Week 52 - central serum | 7900 (NA) — Only one sample analyzed | 203000 (NA) — Only one sample analyzed
  Week 52 - peripheral serum: number analyzed (Participants) | 2 | 2
  Week 52 - peripheral serum | 72000 (37194) | 86510 (122320)
  Week 78 - central serum: number analyzed (Participants) | 0 | 0
  Week 78 - peripheral serum: number analyzed (Participants) | 3 | 2
  Week 78 - peripheral serum | 74450 (105310) | 229500 (101120)
  Week 104 - central serum: number analyzed (Participants) | 1 | 0
  Week 104 - central serum | 79700 (NA) — Only one sample analyzed |
  Week 104 - peripheral serum: number analyzed (Participants) | 2 | 2
  Week 104 - peripheral serum | 292599 (37477) | 195000 (72125)

4. Secondary Outcome: The Time of the End of the Infusion of SOBI003
Description: The time of the end of infusion of SOBI003 (tEnd of inf) Blood samples for serum PK analysis were collected either by centrally (i.e., using a catheter in the central venous port) or peripheral (i.e., by venipuncture). Central venous sampling is more convenient than repeated venipuncture.
Time Frame: Weeks 38, 52, 78 and 104
Population: Number of analysed are available samples
Measure: Median (Full Range); unit: Hours
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
Hours
  Week 38 - central serum: number analyzed (Participants) | 0 | 1
  Week 38 - central serum |  | 6.20 [6.20 to 6.20]
  Week 52 - central serum: number analyzed (Participants) | 1 | 1
  Week 52 - central serum | 4.50 [4.50 to 4.50] | 4.170 [4.17 to 4.17]
  Week 78 - central serum: number analyzed (Participants) | 0 | 0
  Week 104 - central serum: number analyzed (Participants) | 1 | 0
  Week 104 - central serum | 4.47 [4.47 to 4.47] |
  Week 38 - peripheral serum: number analyzed (Participants) | 3 | 2
  Week 38 - peripheral serum | 4.5 [4.08 to 6.25] | 4.825 [4.33 to 5.32]
  Week 52- peripheral serum: number analyzed (Participants) | 2 | 2
  Week 52- peripheral serum | 4.775 [4.08 to 5.47] | 5.845 [4.17 to 7.52]
  Week 78- peripheral serum: number analyzed (Participants) | 3 | 2
  Week 78- peripheral serum | 4.50 [4.18 to 5.88] | 8.575 [4.73 to 12.4]
  Week 104- peripheral serum: number analyzed (Participants) | 2 | 2
  Week 104- peripheral serum | 5.030 [4.03 to 6.03] | 8.540 [4.25 to 12.8]

5. Secondary Outcome: The Maximum Observed Serum Concentration of SOBI003
Description: The maximum observed serum concentration of SOBI003 (Cmax) Blood samples for serum PK analysis were collected either by centrally (i.e., using a catheter in the central venous port) or peripheral (i.e., by venipuncture). Central venous sampling is more convenient than repeated venipuncture.
Time Frame: Weeks 38, 52, 78 and 104
Population: Number of analysed are available samples
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
ng/mL
  Week 38 - central serum: number analyzed (Participants) | 0 | 2
  Week 38 - central serum |  | 105000 [32.0 to 210000]
  Week 52 - central serum: number analyzed (Participants) | 0 | 1
  Week 52 - central serum |  | 203000 [203000 to 203000]
  Week 78 - central serum: number analyzed (Participants) | 1 | 1
  Week 78 - central serum | 136.0 [136.0 to 136.0] | 75.0 [75.0 to 75.0]
  Week 104 - central serum: number analyzed (Participants) | 1 | 0
  Week 104 - central serum | 79700 [79700 to 79700] |
  Week 38 - peripheral serum: number analyzed (Participants) | 3 | 2
  Week 38 - peripheral serum | 7690 [4330 to 31100] | 109500 [107000 to 112000]
  Week 52 - peripheral serum | 45700 [154 to 98300] | 23300 [11600 to 173000]
  Week 78 - peripheral serum: number analyzed (Participants) | 3 | 2
  Week 78 - peripheral serum | 195000 [28000 to 243000] | 229500 [158000 to 301000]
  Week 104 - peripheral serum: number analyzed (Participants) | 2 | 3
  Week 104 - peripheral serum | 292500 [266000 to 319000] | 144000 [25000 to 246000]

6. Secondary Outcome: The Time at Which the Maximum Serum Concentration of SOBI003 is Observed
Description: The time after start of infusion at which the maximum serum concentration is observed (tmax) Blood samples for serum PK analysis were collected either by centrally (i.e., using a catheter in the central venous port) or peripheral (i.e., by venipuncture). Central venous sampling is more convenient than repeated venipuncture.
Time Frame: Weeks 38, 52, 78 and 104
Population: Number of analysed are available samples
Measure: Median (Full Range); unit: Hours
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
Hours
  Week 38 - central serum: number analyzed (Participants) | 0 | 2
  Week 38 - central serum |  | 87.96 [8.17 to 168]
  Week 52 - central serum: number analyzed (Participants) | 1 | 1
  Week 52 - central serum | 4.50 [4.50 to 4.50] | 4.170 [4.170 to 4.170]
  Week 78 - central serum: number analyzed (Participants) | 1 | 1
  Week 78 - central serum | 168 [168 to 168] | 0 [0 to 0]
  Week 104 - central serum: number analyzed (Participants) | 1 | 0
  Week 104 - central serum | 4.47 [4.47 to 4.47] |
  Week 38 - peripheral serum: number analyzed (Participants) | 3 | 2
  Week 38 - peripheral serum | 4.5 [4.08 to 6.25] | 4.825 [4.33 to 5.32]
  Week 52 - peripheral serum | 5.47 [4.08 to 26.5] | 7.52 [0 to 24.5]
  Week 78 - peripheral serum: number analyzed (Participants) | 3 | 2
  Week 78 - peripheral serum | 5.88 [4.5 to 168] | 8.575 [4.73 to 12.4]
  Week 104 - peripheral serum: number analyzed (Participants) | 2 | 3
  Week 104 - peripheral serum | 5.03 [4.03 to 6.03] | 12.83 [4.25 to 23.7]

7. Secondary Outcome: The Minimum Observed Serum Concentration of SOBI003
Description: The minimum observed serum concentration of SOBI003 (CTrough) Blood samples for serum PK analysis were collected either by centrally (i.e., using a catheter in the central venous port) or peripheral (i.e., by venipuncture). Central venous sampling is more convenient than repeated venipuncture.
Time Frame: Weeks 38, 52, 78 and 104
Population: Number of analysed are available samples
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
ng/mL
  Week 38 - central serum: number analyzed (Participants) | 0 | 2
  Week 38 - central serum |  | 68.0 [32.0 to 104.0]
  Week 52 - central serum: number analyzed (Participants) | 0 | 0
  Week 78 - central serum: number analyzed (Participants) | 1 | 1
  Week 78 - central serum | 47.0 [47.0 to 47.0] | 75.0 [75.0 to 75.0]
  Week 104 - central serum: number analyzed (Participants) | 1 | 0
  Week 104 - central serum | 2610 [2610 to 2610] |
  Week 38 - peripheral serum: number analyzed (Participants) | 1 | 2
  Week 38 - peripheral serum | 34 [34 to 34] | 30 [20 to 40]
  Week 52 - peripheral serum: number analyzed (Participants) | 2 | 3
  Week 52 - peripheral serum | 138.5 [123 to 154] | 25 [11 to 45]
  Week 78 - peripheral serum: number analyzed (Participants) | 3 | 1
  Week 78 - peripheral serum | 362 [43 to 28000] | 85 [85 to 85]
  Week 104 - peripheral serum: number analyzed (Participants) | 2 | 3
  Week 104 - peripheral serum | 704.5 [555 to 854] | 75 [13 to 111]

8. Secondary Outcome: Clearance
Description: Clearance (CL) of SOBI003 Blood samples for serum PK analysis were collected either by centrally (i.e., using a catheter in the central venous port) or peripheral (i.e., by venipuncture). Central venous sampling is more convenient than repeated venipuncture.
Time Frame: Weeks 38, 52, 78 and 104
Population: Number of analysed are available samples
Measure: Median (Full Range); unit: mL/min
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
mL/min
  Week 38 - central serum: number analyzed (Participants) | 0 | 0
  Week 52 - central serum: number analyzed (Participants) | 0 | 0
  Week 78 - central serum: number analyzed (Participants) | 1 | 0
  Week 78 - central serum | 208 [208 to 208] |
  Week 104 - central serum: number analyzed (Participants) | 1 | 0
  Week 104 - central serum | 1.6 [1.6 to 1.6] |
  Week 38 - peripheral serum: number analyzed (Participants) | 0 | 1
  Week 38 - peripheral serum |  | 0.661 [0.661 to 0.661]
  Week 52 - peripheral serum: number analyzed (Participants) | 1 | 0
  Week 52 - peripheral serum | 3.51 [3.51 to 3.51] |
  Week 78 - peripheral serum: number analyzed (Participants) | 0 | 0
  Week 104 - peripheral serum: number analyzed (Participants) | 1 | 1
  Week 104 - peripheral serum | 2.21 [2.21 to 2.21] | 3.61 [3.61 to 3.61]

9. Secondary Outcome: Area Under the SOBI003 Serum Concentration-time Curve From Time 0 to168 Hours
Description: Area under the SOBI003 serum concentration-time curve from time 0 to 168 hours (AUC 0-168h) Blood samples for serum PK analysis were collected either by centrally (i.e., using a catheter in the central venous port) or peripheral (i.e., by venipuncture). Central venous sampling is more convenient than repeated venipuncture.
Time Frame: 0,1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168 hours post-dose on Weeks 38, 52, 78 and 104
Population: Number of analysed are available samples
Measure: Median (Full Range); unit: h*ng/mL
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
h*ng/mL
  Week 38 - central serum: number analyzed (Participants) | 0 | 0
  Week 52 - central serum: number analyzed (Participants) | 0 | 0
  Week 78 - central serum: number analyzed (Participants) | 1 | 0
  Week 78 - central serum | 15400 [15400 to 15400] |
  Week 104 - central serum: number analyzed (Participants) | 1 | 0
  Week 104 - central serum | 2040000 [2040000 to 2040000] |
  Week 38 - peripheral serum: number analyzed (Participants) | 0 | 1
  Week 38 - peripheral serum |  | 2880000 [2880000 to 2880000]
  Week 52 - peripheral serum: number analyzed (Participants) | 1 | 0
  Week 52 - peripheral serum | 1110000 [1110000 to 1110000] |
  Week 78 - peripheral serum: number analyzed (Participants) | 0 | 0
  Week 104 - peripheral serum: number analyzed (Participants) | 1 | 1
  Week 104 - peripheral serum | 4390000 [4390000 to 4390000] | 2770000 [2770000 to 2770000]

10. Secondary Outcome: The Half-life
Description: The half-life of SOBI003 in serum (T1/2) Blood samples for serum PK analysis were collected either by centrally (i.e., using a catheter in the central venous port) or peripheral (i.e., by venipuncture). Central venous sampling is more convenient than repeated venipuncture.
Time Frame: Weeks 38, 52, 78 and 104
Population: Number of analysed are available samples
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: SOBI003 Concentration in Cerebrospinal Fluid
Description: Concentration of SOBI003 in cerebrospinal fluid
Time Frame: Weeks 52 and 104
Population: Number analysed are available samples
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
ng/mL
  Week 52: number analyzed (Participants) | 1 | 2
  Week 52 | 15.7 [15.7 to 15.7] | 92.3 [73.6 to 115]
  Week 104: number analyzed (Participants) | 2 | 3
  Week 104 | 118.35 [95.7 to 141.0] | 57.1 [41.5 to 147]

12. Secondary Outcome: Number of Patients Having Anti-drug Antibodies in Serum
Description: Number of patients in each dose group having anti-drug antibodies in serum
Time Frame: Weeks 38, 52, 78 and 104
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
Participants
  Week 38 | 3 | 3
  Week 52 | 3 | 3
  Week 78 | 3 | 2
  Week 104 | 3 | 3

13. Secondary Outcome: Number of Patients Having Anti-drug Antibodies in Cerebrospinal Fluid
Description: Number of patients in each dose group having anti-drug antibodies cerebrospinal fluid
Time Frame: Weeks 52 and 104
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
Participants
  Week 52 | 2 | 3
  Week 104 | 3 | 3

14. Secondary Outcome: Change From Baseline in Heparan Sulfate Concentration in Cerebrospinal Fluid
Description: Change from baseline, in percent, of Heparan Sulfate levels in cerebrospinal fluid
Time Frame: Weeks 52 and 104
Measure: Median (Full Range); unit: mg/L
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
mg/L
  Week 52 | -1.19 [-4.91 to 0.1] | -3.47 [-23.2 to -2.579]
  Week 104 | -6.07 [-6.67 to -4.42] | -3.59 [-24.7 to -2.18]

15. Secondary Outcome: Change From Baseline in Heparan Sulfate Levels in Serum
Description: Change from baseline in Heparan sulfate, in mg/L, levels in serum
Time Frame: Weeks 38, 52, 78 and 104
Measure: Median (Full Range); unit: mg/L
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
mg/L
  Week 38 | -1.811 [-2.168 to -1.793] | -1.88 [-3.721 to -1.854]
  Week 52 | -1.76 [-2.169 to -1.644] | -2.25 [-3.735 to -1.18]
  Week 78 | -1.729 [-2.41 to -1.686] | -2.01 [-3.05 to -0.97]
  Week 104 | -2.21 [-2.41 to 0.21] | -2.24 [-3.708 to -1.91]

16. Secondary Outcome: Change From Baseline in Heparan Sulfate Levels in Urine
Description: Change from baseline in Heparan sulfate levels, in g/mol, in urine
Time Frame: Weeks 38, 52, 78 and 104
Population: Number of analysed are available samples
Measure: Median (Full Range); unit: g/mol
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
g/mol
  Week 38 | -447.2 [-552.82 to -340.1] | -692.78 [-697.12 to -382.65]
  Week 52 | -464.4 [-559.02 to -411.67] | -698.79 [-701.99 to -388.86]
  Week 78: number analyzed (Participants) | 2 | 2
  Week 78 | -512.19 [-599.70 to -424.68] | -494.610 [-747.22 to -242.0]
  Week 104 | -578.89 [-709.47 to -489.68] | -726.24 [-753.97 to -381.45]

17. Secondary Outcome: Change From Baseline in Neurocognitive Development Quotient
Description: Quotient between age equivalent score and age, 0 - 100%, where high values are desirable. The age equivalent score represent the age of the typical and normal individual who would achieve the same result as the one who was tested The age equivalent scores are assessed by the Bayley Scales of Infant and Toddler Development®, third edition cognitive subtest or the Kaufman Assessment Battery for Children, Second edition.
  The Bayley Scales of Infant and Toddler Development-Third Edition is an individually administered test designed to assess developmental functioning of infants and toddlers. The Bayley-III assesses development in five areas: cognitive, language, motor,social-emotional, and adaptive behavior.
  The Kaufman Assessment Battery for Children (K-ABC) is a clinical instrument for assessing cognitive development.
  These results are truly "unitless"/"dimensionless" because they represents quotients of values from the same scale, which means that the units in the denominator and
Time Frame: Weeks 52 and 104
Population: Number of analysed are number of assessments
Measure: Median (Full Range); unit: Unitless
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
Unitless
  Week 52: number analyzed (Participants) | 3 | 2
  Week 52 | -8.97 [-18 to -6.9] | -31.74 [-48.9 to -14.6]
  Week 104 | -16.28 [-32.9 to -11.7] | -24.94 [-44.6 to -11.3]

18. Secondary Outcome: Change From Baseline in Age-equivalence Score
Description: The age equivalent score represent the age in months of the typical and normal individual who would achieve the same result as the one who was tested. The age equivalent scores are assessed by the Bayley Scales of Infant and Toddler Development®, third edition cognitive subtest or the Kaufman Assessment Battery for Children, Second edition. The Bayley Scales of Infant and Toddler Development-Third Edition is an individually administered test designed to assess developmental functioning of infants and toddlers. The Bayley-III assesses development in five areas: cognitive, language, motor, social-emotional, and adaptive behavior. The Kaufman Assessment Battery for Children (K-ABC) is a clinical instrument for assessing cognitive development.
Time Frame: Week 52 and 104
Population: Number of analyses are available assessments
Measure: Median (Full Range); unit: Months
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
Months
  Week 52: number analyzed (Participants) | 3 | 2
  Week 52 | -1.0 [-2 to 2] | -1.0 [-2 to 0]
  Week 104 | -3.0 [-4 to 1] | 5.0 [-1 to 10]

19. Secondary Outcome: Age-equivalence Score as Assessed Either by the BSID-III, Cognitive Subtest, or the KABC-II.
Description: The age equivalent score represent the age in months of the typical and normal individual who would achieve the same result as the one who was tested. The age equivalent scores are assessed by Vineland™ Adaptive Behavior Scales, Expanded Interview Form, Second edition (VABS-II). The Vineland is designed to measure adaptive behavior of individuals from birth to age 90. The Vineland-II contains 5 domains each with 2-3 subdomains. The main domains are: Communication, Daily Living Skills, Socialization, Motor Skills, and Maladaptive Behavior.
Time Frame: Week 52 and 104
Population: Number of analyses are available assessments
Measure: Median (Full Range); unit: Months
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
Months
  Week 52: number analyzed (Participants) | 3 | 2
  Week 52 | 14.0 [10 to 31] | 16.0 [12 to 20]
  Week 104 | 13.0 [8 to 29] | 19.0 [19 to 36]

20. Secondary Outcome: Change From Baseline in Age-equivalence Score as Assessed Either by the BSID-III, Cognitive Subtest, or the KABC-II.
Description: The age equivalent score represents the age in months of the typical and normal individual who would achieve the same result as the one who was tested.
  The age equivalent scores are assessed either by the Bayley Scales of Infant and Toddler Development®, third edition, (BSID-III) cognitive subtest or the Kaufman Assessment Battery for Children, Second edition (KABC-II) depending on chronological age of the subject. Quotient between age equivalent score and age, 0 - 100%, where high values are desirable.
  The BSID-III is an individually administered test designed to assess developmental functioning of infants and toddlers. The BSID-III assesses development in five areas: cognitive, language, motor, social-emotional, and adaptive behavior.
  The KABC-II is a clinical instrument for assessing cognitive development. The unit and measurement is the same in both scales (BSID-III and KABC-II): Age-equivalent score.
Time Frame: Week 52 and 104
Population: Number of analysed are available assessments
Measure: Median (Full Range); unit: Months
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
Months
  Week 52: number analyzed (Participants) | 3 | 2
  Week 52 | -1.0 [-2 to 2] | -1.0 [-2 to 0]
  Week 104 | -3.0 [-4 to 1] | 5.0 [-1 to 10]

21. Secondary Outcome: Age-equivalence Score as Assessed by VABS-II
Description: as for outcome 19
Time Frame: Week 52 and 104
Measure: Median (Full Range); unit: Months
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
Months
  Week 52 | 15 [15 to 26] | 28 [13 to 37]
  Week 104 | 16 [13 to 21] | 23 [20 to 43]

22. Secondary Outcome: Change From Baseline in Age-equivalence Score as Assessed by VABS-II
Description: as for outcome 19
Time Frame: Week 52 and 104
Measure: Median (Full Range); unit: Months
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
Months
  Week 52 | -1 [-12 to 2] | 1 [0 to 4]
  Week 104 | -6 [-11 to 0] | 8 [-5 to 10]

23. Secondary Outcome: Change From Baseline in Gray Matter Volume
Description: Grey matter contains most of the brain's neuronal cell bodies. The grey matter includes regions of the brain involved in muscle control, and sensory perception such as seeing and hearing, memory, emotions, speech, decision making, and self-control. The gray matter volume will be measured by volumetric magnetic resonance imaging (MRI) at weeks 52 and 104.
Time Frame: Week 52 and 104
Population: Number analysed is available assessments
Measure: Median (Full Range); unit: mL
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
mL
  Week 52: number analyzed (Participants) | 3 | 2
  Week 52 | -24.629 [-34.32 to 66.87] | 19.485 [-62.32 to 101.29]
  Week 104: number analyzed (Participants) | 2 | 2
  Week 104 | -53.584 [-161.03 to 53.86] | 13.387 [-45.41 to 72.18]

24. Secondary Outcome: Pediatric Quality of Life Inventory (PedsQL™) Total Score
Description: Pediatric Quality of Life Inventory (PedsQL™) is a modular approach to measuring health-related quality of life in healthy children and adolescents and those with acute and chronic health conditions. Lower scores indicate better functioning. Min score = 0, and max score = 144.
Time Frame: Week 52 and 104
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
Units on a scale
  Week 52 | 53.4 (3.9) | 72.2 (11.6)
  Week 104 | 55.9 (10.2) | 76.5 (3.8)

25. Secondary Outcome: Change From Baseline in Pediatric Quality of Life Inventory (PedsQL™) Total Score
Description: Pediatric Quality of Life Inventory (PedsQL™) is a modular approach to measuring health-related quality of life (HRQOL) in healthy children and adolescents and those with acute and chronic health conditions. Higher scores indicate better functioning. Min score = 0, and max score = 144.
Time Frame: Week 52 and 104
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
Units on a scale
  Week 52 | -17.0 (25.9) | -3.7 (24.2)
  Week 104 | -14.5 (14.9) | 0.6 (21.0)

26. Secondary Outcome: PedsQL™ Family Impact Module Total Score
Description: Pediatric Quality of Life Inventory (PedsQL™) is a modular approach to measuring health-related quality of life in healthy children and adolescents and those with acute and chronic health conditions. The Total Score is the sum of all 36 items in the test divided by the number of items answered. Higher scores indicate better functioning. Min score = 0, and max score = 144.
Time Frame: Week 52 and 104
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
Units on a scale
  Week 52 | 66.7 (30.6) | 70.0 (26.5)
  Week 104 | 73.3 (34.0) | 70.0 (26.5)

27. Secondary Outcome: Change From Baseline in PedsQL™ Family Impact Module Total Score
Description: Pediatric Quality of Life Inventory (PedsQL™) is a modular approach to measuring health-related quality of life in healthy children and adolescents and those with acute and chronic health conditions. The Total Score is the sum of all 36 items in the test divided by the number of items answered. Higher scores indicate better functioning.
Time Frame: Week 52 and 104
Population: Number analysed is available assessments
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
Units on a scale
  Week 52: number analyzed (Participants) | 3 | 2
  Week 52 | 16.7 (12.6) | 0.0 (0.0)
  Week 104: number analyzed (Participants) | 3 | 2
  Week 104 | 23.3 (31.8) | 0.0 (0.0)

ADVERSE EVENTS:
Time Frame: The period for recording adverse events, including Serious Adverse Events (SAEs), began Day 1 of week 25, when first dose in study SOBI003-002 was given, and ended at completion of week 104 visit. In addition SAEs was reported from the time of signing the informed consent form until 28 days past the last dose of SOBI003.
Arm/Group | Dose Group 1 | Dose Group 2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Group 1 (N=3) | Dose Group 2 (N=3)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (2)
Device related infection (Infections and infestations) | 0 | 1 (1)
Endocarditis (Infections and infestations) | 0 | 1 (1)
Infection (Infections and infestations) | 0 | 1 (1)
Influenza (Infections and infestations) | 0 | 1 (1)
Pneumonia (Infections and infestations) | 0 | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 | 1 (1)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Group 1 (N=3) | Dose Group 2 (N=3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (2) | 1 (2)
Aortic valve thickening (Cardiac disorders) | 0 (0) | 1 (1)
Cyanosis (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (20) | 3 (28)
Auricular swelling (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Otorrhoea (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (4) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (10)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (4)
Oral contusion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (17) | 3 (22)
Application site erythema (General disorders) | 0 (0) | 1 (1)
Catheter site extravasation (General disorders) | 0 (0) | 1 (1)
Catheter site inflammation (General disorders) | 1 (1) | 1 (1)
Catheter site injury (General disorders) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 1 (6)
Fatigue (General disorders) | 0 (0) | 1 (1)
Infusion site bruising (General disorders) | 1 (1) | 0 (0)
Infusion site irritation (General disorders) | 0 (0) | 1 (1)
Medical device site haemorrhage (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (8) | 3 (11)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (2) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (2) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (4) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (17) | 2 (12)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (2) | 3 (8)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 1 (8)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Human bite (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 1 (6)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (10)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (4)
Vascular access site occlusion (Injury, poisoning and procedural complications) | 1 (4) | 2 (5)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (3)
Blood fibrinogen increased (Investigations) | 0 (0) | 1 (2)
Blood pressure diastolic increased (Investigations) | 0 (0) | 1 (1)
Blood pressure systolic increased (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (2)
CSF glucose decreased (Investigations) | 0 (0) | 1 (1)
CSF protein increased (Investigations) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 0 (0) | 1 (1)
Eosinophil count increased (Investigations) | 0 (0) | 1 (2)
Haemoglobin increased (Investigations) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 1 (1)
Monocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 2 (26)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Red blood cell count increased (Investigations) | 0 (0) | 1 (1)
Vitamin D decreased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (2)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Clonus (Nervous system disorders) | 0 (0) | 1 (2)
Drooling (Nervous system disorders) | 0 (0) | 1 (2)
Tremor (Nervous system disorders) | 1 (1) | 2 (6)
Device damage (Product Issues) | 1 (2) | 0 (0)
Device dislocation (Product Issues) | 1 (2) | 2 (2)
Device malfunction (Product Issues) | 1 (1) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 2 (8)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (10)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (22)
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (7)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (13) | 2 (4)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (13)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (20) | 3 (20)
Flushing (Vascular disorders) | 0 (0) | 3 (5)
Hyperaemia (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-06-29): https://cdn.clinicaltrials.gov/large-docs/28/NCT03811028/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-13): https://cdn.clinicaltrials.gov/large-docs/28/NCT03811028/SAP_001.pdf